CLINICAL TRIAL: NCT00783679
Title: Determining the Feasibility and Accuracy of Exhaled CO2 to Measure Cardiac Output in Ventilated Patients Without Tracheal Intubation
Brief Title: The Feasibility and Accuracy of Exhaled CO2 to Measure Cardiac Output in Ventilated Patients Without Tracheal Intubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Understaffing and inadequate funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Professor of Anesthesia, Director of Respiratory Care Services, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2007-P-000222
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Cardiac Physiology; Cardiac Output
Keywords: Cardiac output; Noninvasive cardiac output measurement; Thermodilution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Twenty adult spontaneously breathing patients without intubation and mechanical ventilation recruited from the cardiac catheterization laboratory. All will be post-heart-transplant patients coming for yearly evaluation.
  Interventions: Device: NICO device

INTERVENTIONS:
Device: NICO device — Measurement of cardiac output and simultaneous blood sampling.
  The subjects' cardiac output will be measured by NICO device and also by thermodilution method. Simultaneously blood samples will be drawn from the pulmonary artery catheter and arterial line. The calculated and measured cardiac output values will be compared for accuracy.

SUMMARY:
The purpose of this study is to test the accuracy of a new noninvasive way to measure how much blood our heart pumps per minute. This new way measures the heart's pumping activity from outside the body, instead of breaking the skin and measuring it from the inside.

Subjects will breathe normally through a mask while we record how fast and how much air they are breathing. We will have them "re-breathe" some of the air they breathed out by adjusting the ventilator. During this time, we will use the air breathed out to calculate how much blood per minute the subject's heart is pumping. We will also measure how much blood the heart is pumping at this time by injecting fluid into the catheter in the neck and then drawing about 1 teaspoon of blood from the catheters in the neck and arm. We will compare the calculated and measured values of the amount of blood pumped out of the heart for accuracy.

After we complete this procedure, we will remove the mask and allow you to rest for 10-30min. Following the rest period, we will repeat the process and collect a second set of measurements. We will draw a total of 4 teaspoons of blood for the study.

If you cannot comfortably breathe along with the ventilator, we will withdraw you from the study. If you want to stop taking part in the study at any time, let the study doctor know that you wish to withdraw. We will take off the mask, and your time in the study will end. This decision will not affect your regular medical care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is already monitored with a pulmonary artery catheter and arterial line (not for the purpose of this study);
2. Hemodynamic stability.

Exclusion Criteria:

1. Patients with facial deformity, heavy beard or moustache which prevents good seal between the mask and the face;
2. Patients who have central nervous system disorders that might be adversely affected by CO2 rebreathing, such as head trauma patients with increased intracranial pressure;
3. Patients with severe tricuspid regurgitation;
4. Patients with intra-cardiac shunts;
5. Patients who cannot cooperate and synchronize with the ventilator;
6. Patients with unstable respiratory conditions, such as acute respiratory failure;
7. Patients who have claustrophobia and cannot wear the mask.
8. Patients with aortic stenosis.
9. Patients with left main coronary artery disease.
10. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To test the feasibility and accuracy of using NICO to measure cardiac output in ventilator assisted patients without tracheal intubation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, PhD, RRT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States